CLINICAL TRIAL: NCT02066116
Title: Effect of Kinect-based Upper Limb Rehabilitation System in Patients With Stroke: A Pilot Trial
Brief Title: Kinect-based Upper Limb Rehabilitation System in Stroke Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment is difficult and pilot nature of this study
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Microsoft Research (Industry); Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Nam-Jong Paik, MD, PhD, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1401-234-001
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Stroke; Hemiplegia; Virtual Rehabilitation
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinect-based Rehabilitation (Experimental)
  Interventions: Procedure: Kinect-based rehabilitation plus occupational therapy
- Self-exercises education (Active Comparator)
  Interventions: Other: sham virtual rehabilitation education plus occupational therapy

INTERVENTIONS:
Procedure: Kinect-based rehabilitation plus occupational therapy — The developed kinect-based rehabilitation system will be used for 30min/session. Conventional 30min occupational therapy also will be applied for the patient enrolled.
  Arms: Kinect-based Rehabilitation
Other: sham virtual rehabilitation education plus occupational therapy — For the sham virtual rehabilitation, computer-based cognitive rehabilitation program will be used. Patients will be encouraged to use their affected arm to push the button but the motion will be minimal and not related to the concept of upper extremity rehabilitation.
  Arms: Self-exercises education

SUMMARY:
The investigators have developed the kinect-based upper extremity rehabilitation program and designed this protocol to prove the efficacy of this program.

In brief, subacute stroke patients allocated to intervention group will receive the kinect based-rehabilitation program plus conventional occupational therapy and patients allocated to control group will receive the sham virtual rehabilitation plus conventional occupational therapy, for 10 days.

20 patients with subacute stroke will be allocated into each group and after completing the 10 days intervention, they will be assessed by using objective assessment tools for upper extremity function.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 80 years
* Stroke within prior 3 months
* Unilateral upper extremity weakness

Exclusion Criteria:

* Uncontrolled medical conditions
* Who cannot obey the simple command
* Who has the hemispatial neglect, visual impairment, apraxia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Fugl-Meyer Assessment Scale for upper extremity at 2 weeks | Baseline, 2 weeks after the baseline

SECONDARY OUTCOMES:
Brunnstrom stage | Baseline, 2 weeks after the baseline, 6 weeks after the baseline, 14 weeks after the baseline
  This is composed of 6 stages. Higher score means better function. The description for each stage as follows.
  1. Flaccidity: no voluntary movement.
  2. Synergies or minimal voluntary movement.
  3. Synergies performed voluntary (spasticity gratest).
  4. Some deviation from synergy.
  5. Independent or isolated movement.
  6. Individual joint movement nearly normal with minimal spasticity.
Modified Barthel Index | Baseline, 2 weeks after the baseline, 6 weeks after the baseline, 14 weeks after the baseline
Box and Block Test | Baseline, 2 weeks after the baseline, 6 weeks after the baseline, 14 weeks after the baseline
  Individuals are seated at a table, facing a rectangular box that is divided into two square compartments of equal dimension by means of a partition.
  One hundred and fifty, 2.5 cm, colored, wooden cubes or blocks are placed in one compartment or the other.
  The individual is instructed to move as many blocks as possible, one at a time, from one compartment to the other for a period of 60 seconds.
  The BBT is scored by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period.
Number of movement counts during rehabilitation using accelerometer data | Baseline, 2 weeks after the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam, Korea
Locations (1):
- Seoul National University Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://research.microsoft.com/en-us/default.aspx
- See also: Related Info — http://www.youtube.com/watch?v=PVgiEtDbsQM#t=15